CLINICAL TRIAL: NCT04986930
Title: Randomized Phase 2 Study of mFOLFIRINOX With or Without Stereotactic Body Radiotherapy in Patients With Locally Advanced Pancreatic Adenocarcinoma
Brief Title: mFOLFIRINOX With or Without Stereotactic Body Radiotherapy in Locally Advanced Pancreatic Adenocarcinoma
Acronym: SABER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Changhoon Yoo, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SABER
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Cancer Non-resectable
Keywords: Pancreatic adenocarcinoma; Locally advanced unresectable; mFOLFIRINOX; Stereotactic body radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SBRT+mFOLFIRINOX (Experimental): * Stereotactic body radiotherapy: 3500 cGy (5 fractions)
  * mFOLFIRINOX, every 2 weeks Oxaliplatin, 85 mg/m2, intravenous, day 1 Leucovorin, 400 mg/m2, intravenous, day 1 Irinotecan, 150 mg/m2, intravenous, day 1 fluorouracil, 2,400 mg/m2, intravenous, day 1-2
  Interventions: Radiation: SBRT+mFOLFIRINOX
- mFOLFIRINOX (Active Comparator): -mFOLFIRINOX, every 2 weeks Oxaliplatin, 85 mg/m2, intravenous, day 1 Leucovorin, 400 mg/m2, intravenous, day 1 Irinotecan, 150 mg/m2, intravenous, day 1 fluorouracil, 2,400 mg/m2, intravenous, day 1-2
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Radiation: SBRT+mFOLFIRINOX — Stereotactic body radiotherapy: 3500 cGy (5 fractions) mFOLFIRINOX, every 2 weeks Oxaliplatin, 85 mg/m2, intravenous, day 1 Leucovorin, 400 mg/m2, intravenous, day 1 Irinotecan, 150 mg/m2, intravenous, day 1 fluorouracil, 2,400 mg/m2, intravenous, day 1-2
  Arms: SBRT+mFOLFIRINOX
Drug: mFOLFIRINOX — mFOLFIRINOX, every 2 weeks Oxaliplatin, 85 mg/m2, intravenous, day 1 Leucovorin, 400 mg/m2, intravenous, day 1 Irinotecan, 150 mg/m2, intravenous, day 1 fluorouracil, 2,400 mg/m2, intravenous, day 1-2
  Arms: mFOLFIRINOX

SUMMARY:
Modified FOLFIRINOX (mFOLFIRINOX) is the standard of care for patients with locally advanced pancreatic adenocarcinoma. While radiotherapy has been investigated for the management of resectable or locally advanced pancreatic adenocarcinoma, its role in the era of modern chemotherapy is not clear. Stereotactic body radiotherapy (SBRT) is the novel technique of radiotherapy to enhance the dose of radiotherapy to the target tumor lesion. This trial aims to compare the efficacy and safety of mFOLFIRINOX with or without SBRT in patients with locally advanced pancreatic adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 19 years or greater
* Cytologically or histologically confirmed pancreatic adenocarcinoma
* Locally advanced unresectable disease per National Comprehensive Cancer Network resectability criteria
* No active infection except chronic hepatitis on anti-viral therapy
* Eastern Cooperative Oncology Group performance status 0 or 1
* Body weight > 30 kg
* Normal organ and bone marrow function

Exclusion Criteria:

* Gastrointestinal obstruction
* Active gastrointestinal bleeding or ulcer
* Clinically significant cardiac disease or myocardial infarction within 6 months before the randomization
* Histology other than adenocarcinoma (adenosquamous or neuroendocrine tumors)
* Pregnancy or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-08-14 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-12-14 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival rate | 1 year
  Proportion of patients without disease progression or death

SECONDARY OUTCOMES:
Overall survival | 1 year
  Time between randomization and death of any cause
Progression-free survival | 1 year
  Time between randomization and disease progression or death of any cause
Overall response rates | 1 year
  Tumor response per Response Evaluation Criteria in Solid Tumors version 1.1
Adverse events | 1 year
  Any unintended events graded per National Cancer Institute Common Terminology Criteria for Adverse Events version 5
Surgical resection rate | 1 year
  Proportion of patients who underwent curative-intent surgery

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balaban EP, Mangu PB, Khorana AA, Shah MA, Mukherjee S, Crane CH, Javle MM, Eads JR, Allen P, Ko AH, Engebretson A, Herman JM, Strickler JH, Benson AB 3rd, Urba S, Yee NS. Locally Advanced, Unresectable Pancreatic Cancer: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2016 Aug 1;34(22):2654-68. doi: 10.1200/JCO.2016.67.5561. Epub 2016 May 31. PMID 27247216
- [Background] Hammel P, Huguet F, van Laethem JL, Goldstein D, Glimelius B, Artru P, Borbath I, Bouche O, Shannon J, Andre T, Mineur L, Chibaudel B, Bonnetain F, Louvet C; LAP07 Trial Group. Effect of Chemoradiotherapy vs Chemotherapy on Survival in Patients With Locally Advanced Pancreatic Cancer Controlled After 4 Months of Gemcitabine With or Without Erlotinib: The LAP07 Randomized Clinical Trial. JAMA. 2016 May 3;315(17):1844-53. doi: 10.1001/jama.2016.4324. PMID 27139057
- [Background] Loehrer PJ Sr, Feng Y, Cardenes H, Wagner L, Brell JM, Cella D, Flynn P, Ramanathan RK, Crane CH, Alberts SR, Benson AB 3rd. Gemcitabine alone versus gemcitabine plus radiotherapy in patients with locally advanced pancreatic cancer: an Eastern Cooperative Oncology Group trial. J Clin Oncol. 2011 Nov 1;29(31):4105-12. doi: 10.1200/JCO.2011.34.8904. Epub 2011 Oct 3. PMID 21969502
- [Background] Murphy JE, Wo JY, Ryan DP, Jiang W, Yeap BY, Drapek LC, Blaszkowsky LS, Kwak EL, Allen JN, Clark JW, Faris JE, Zhu AX, Goyal L, Lillemoe KD, DeLaney TF, Fernandez-Del Castillo C, Ferrone CR, Hong TS. Total Neoadjuvant Therapy With FOLFIRINOX Followed by Individualized Chemoradiotherapy for Borderline Resectable Pancreatic Adenocarcinoma: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Jul 1;4(7):963-969. doi: 10.1001/jamaoncol.2018.0329. PMID 29800971